CLINICAL TRIAL: NCT05969210
Title: Effects of Big Toe Strengthening on Agility, Jump and Speed Among Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0423 Aqsa
Record Dates: First submitted 2023-06-06; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Sports Physical Therapy
Keywords: Big toe; Athlete; Dynamometer; Muscle Strength; Agility
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 12 participants will be in experimental group giving them Toe strengthening exercise protocol along with running training for three weeks, measure all values before giving them protocol and after protocol.
  Interventions: Other: Toe strengthening exercise
- Group B (Experimental): 12 participants will be in control group they will do only there running training.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Toe strengthening exercise — 12 participants will be in experimental group giving them Toe strengthening exercise protocol along with running training for three weeks, measure all values before giving them protocol and after protocol.
  Arms: Group A
Other: Control Group — 12 participants will be in control group they will do only there running training.
  Arms: Group B

SUMMARY:
Running form and technique have a direct influence on a runner's economy, and therefore small changes in specific running mechanics could be useful to improving running performance. The thumb plays an important role in the functionality of the foot. During standing, the big toe is more loaded than the head of the five metatarsals and the heel.

The study design will be a Randomized Controlled Trial. This study will be conducted in Pakistan Sports Board (PSB) Lahore. The study will be completed within the time duration of eight to ten months after the approval of the synopsis. The sample size will be 30 subjects. Non-probability convenient sampling technique will be used to recruit the individuals for the study. Then randomization will be done by lottery method to divide the individuals into 2 treatment groups. The experimental group is given big toe strengthening program for 3 weeks along with running training on the other hand control group will do only their running training and after that measure their pre-post values on spss.

In this study, it will be aimed to examine the relationship of big toe strength with parameters that affect anaerobic athletic performance in runners such as vertical jump, horizontally jumping, strength, agility and speed.

DETAILED DESCRIPTION:
The objective of my study is to explore the effects of big toe strengthening on agility, jump and speed among runners.

ELIGIBILITY:
Inclusion Criteria:

* Age; 16-28yrs
* Male runners
* Doing Running practice for 3 days in a week(40-60minutes per day)

Exclusion Criteria:

* Participants a will be excluded if they have any neurological signs.
* Any lower limb trauma and history of fracture past six month
* Systematic illness ; diabetic ,hypertension(6)

Ages: 16 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
HIP AND TOE DYNAMOMETER | 3 weeks
  Athletes will placed their feet on the ground prepared in accordance with the big toe and adjusted their big toes according to the location of the pinch meter. During the measurement, athletes will asked to apply maximum force with their big toe. Strength measurements were made on the athletes in the sitting position without any support(6).
Dynamic balance Y TEST, Star excursion test (SEBT) | 3 weeks
  Y test reliability (ICC = 0.88- 0.99 (14) The reliability of the SEBT as being moderate to good (ICC 0.67- 0.97 )(14).
Vertical jumping, Horizontal jumping | 3 weeks
  puts chalk on their fingertips to mark the wall at the height of their jump. Then stands away from the wall, and jumps vertically as high as possible using both arms and legs to assist in projecting the body upwards. Attempt to touch the wall at the highest point of the jump(15)
STRENGHT • Speed: 20m Sprint test • Agility---- T- Test | 3 weeks
  Ask the player to put the thumb on dynamometer and press it and see the strength.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denadai BS, Greco CC. Could middle- and long-distance running performance of well-trained athletes be best predicted by the same aerobic parameters? Curr Res Physiol. 2022 Jun 23;5:265-269. doi: 10.1016/j.crphys.2022.06.006. eCollection 2022. PMID 35800136
- [Background] Tufano JJ, Amonette WE. Assisted versus resisted training: which is better for increasing jumping and sprinting? Strength & Conditioning Journal. 2018;40(1):106-10.
- [Background] Horicka P, Simonek J, Brodani J. Diagnostics of reactive and running agility in young football players. Physical Activity Review. 2018;6:29-36.
- [Background] Stoneham R, Barry G, Saxby L, Wilkinson M. The influence of great toe valgus on pronation and frontal plane knee motion during running. The Foot and Ankle Online Journal. 2020;13(1):7.
- [Background] Angin S, Demirbüken İ. Ankle and foot complex. Comparative Kinesiology of the Human Body: Elsevier; 2020. p. 411-39.
- [Background] Sarikaya F, Sahin M. The Effect of Big Toe Strength Development on Some Athletic Performance Parameter in Young Male Footballers. Pakistan Journal of Medical & Health Sciences. 2022;16(02):997-.
- [Background] Kurihara T, Terada M, Numasawa S, Kusagawa Y, Maeo S, Kanehisa H, Isaka T. Effects of age and sex on association between toe muscular strength and vertical jump performance in adolescent populations. PLoS One. 2021 Dec 31;16(12):e0262100. doi: 10.1371/journal.pone.0262100. eCollection 2021. PMID 34972181
- [Background] Sutkowska E, Sutkowski K, Sokolowski M, Franek E, Dragan S Sr. Distribution of the Highest Plantar Pressure Regions in Patients with Diabetes and Its Association with Peripheral Neuropathy, Gender, Age, and BMI: One Centre Study. J Diabetes Res. 2019 Jul 9;2019:7395769. doi: 10.1155/2019/7395769. eCollection 2019. PMID 31380446
- [Background] Liang ZQ, Meng Y, Popik S, Chen FF, editors. Analysis of foot morphology in habitually barefoot group. Journal of Biomimetics, Biomaterials and Biomedical Engineering; 2019: Trans Tech Publ.
- [Background] Yamauchi J, Koyama K. The mechanical role of the metatarsophalangeal joint in human jumping. PLoS One. 2022 May 20;17(5):e0268634. doi: 10.1371/journal.pone.0268634. eCollection 2022. PMID 35594285
- [Background] Yamauchi J, Koyama K. Importance of toe flexor strength in vertical jump performance. J Biomech. 2020 May 7;104:109719. doi: 10.1016/j.jbiomech.2020.109719. Epub 2020 Feb 26. PMID 32173032
- [Background] Otsuka M, Yamauchi J, Kurihara T, Morita N, Isaka T. Toe flexor strength and lower-limb physical performance in adolescent. Gazzetta medica italiana. 2015;174(7-8):307-13.
- [Background] Shin H, Moon SW, Kim GS, Park JD, Kim JH, Jung MJ, Yoon CH, Lee ES, Oh MK. Reliability of the pinch strength with digitalized pinch dynamometer. Ann Rehabil Med. 2012 Jun;36(3):394-9. doi: 10.5535/arm.2012.36.3.394. Epub 2012 Jun 30. PMID 22837976
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Young W, Wilson G, Byrne C. Relationship between strength qualities and performance in standing and run-up vertical jumps. J Sports Med Phys Fitness. 1999 Dec;39(4):285-93. PMID 10726428
- [Background] Dobbs CW, Gill ND, Smart DJ, McGuigan MR. Relationship between vertical and horizontal jump variables and muscular performance in athletes. J Strength Cond Res. 2015 Mar;29(3):661-71. doi: 10.1519/JSC.0000000000000694. PMID 25226312
- [Background] Pauole K, Madole K, Garhammer J, Lacourse M, Rozenek R. Reliability and validity of the T-test as a measure of agility, leg power, and leg speed in college-aged men and women. The Journal of Strength & Conditioning Research. 2000;14(4):443-50.